CLINICAL TRIAL: NCT05722561
Title: Effectiveness and Impact of Counseling Enhanced With Electronic Cigarettes for Harm Reduction in Smokers With Opioid Use Disorder
Brief Title: E-Cigarettes for Harm Reduction in Smokers With Opioid Use Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-00661
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Opioid Use Disorder; Cigarette Smoking
Keywords: cigarettes; smoking; smoking reduction; OUD; OUDTP; Buprenorphine; Methadone
MeSH Terms: conditions — Opioid-Related Disorders; Cigarette Smoking; Smoking; Smoking Reduction | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Electronic Cigarette (Experimental): Participants in the Electronic Cigarette (EC) arm will receive telehealth motivational counseling for 5 weeks plus the standardized research e-cigarette (SREC).
  Interventions: Behavioral: Telehealth Motivational Counseling; Device: National Institute on Drug Abuse (NIDA) Standardized Research Electronic Cigarette (SREC).
- Nicotine Replacement Therapy (Active Comparator): Participants in the Nicotine Replacement Therapy (NRT) arm will receive telehealth motivational counseling plus combination NRT (patch and lozenge).
  Interventions: Behavioral: Telehealth Motivational Counseling; Drug: Nicotine Replacement Product

INTERVENTIONS:
Behavioral: Telehealth Motivational Counseling — At baseline, after randomization, participants will receive their first telehealth session (20~25 minutes) from a counselor trained in motivational interviewing, harm reduction, and smoking cessation. Four additional sessions will be delivered (weeks 2, 3, 4, 6), 15~20 minutes each.
Drug: Nicotine Replacement Product — Combination nicotine replacement therapy with lozenges and patches. Participants are recommended to use the NRT according to product directions.
  Arms: Nicotine Replacement Therapy
Device: National Institute on Drug Abuse (NIDA) Standardized Research Electronic Cigarette (SREC). — Participants are to use the electronic cigarette freely as replacement for smoking combustible cigarettes.
  Arms: Electronic Cigarette

SUMMARY:
The purpose of this an open-label, randomized controlled trial study is to compare the effectiveness of electronic cigarettes (e-cigarettes/e-cigs) versus telehealth motivational counseling with combination nicotine replacement therapy (NRT) + telehealth counseling on combustible cigarettes smoking reduction among persons with opioid use disorder (OUD) in methadone and buprenorphine treatment programs (opioid use disorder treatment programs (OUDTP)). OUDTP patients are a population with exceptionally high combustible cigarettes smoking burden and yet limited success in achieving meaningful clinical outcomes in tobacco treatment. If effective, electronic cigarettes would provide an additional tool for tobacco harm reduction among this difficult-to-treat vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

1. Currently smokes 5 or more CPD
2. Age ≥ 21 years
3. Has a diagnosis of Opioid Use Disorder
4. In OUDTP (buprenorphine or methadone) ≥ 12 weeks via self-report or EHR records
5. Stable methadone or buprenorphine dose for two weeks via self-report or EHR records
6. Interested in reducing combustible cigarette (CC) smoking but not necessarily trying to quit
7. Own a mobile phone or have regular access to a mobile phone.
8. Able to provide an additional contact to improve follow-up rates.

Exclusion Criteria:

1. Does not speak English or Spanish
2. Are pregnant or breastfeeding
3. Not able to provide consent
4. Used tobacco products other than CC in the past 2 weeks (e.g., EC, cigarillo)
5. Currently engaged in an attempt to quit CC smoking
6. Reports having severe chronic obstructive pulmonary disease or asthma (i.e., with exacerbation requiring hospitalization or intubation in the prior 6 months)
7. Reports current major depressive or manic episode, current psychotic disorder, past-year suicide attempt or psychiatric hospitalization, or current suicidal ideation with plan or intent.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve 100% Reduction in Cigarettes Per Day (CPD) between Baseline and End of Intervention (Visit 5) | Up to Visit 5 (Day 56)
  Verified by exhaled carbon-monoxide (eCO) level.

SECONDARY OUTCOMES:
Percentage of Participants who Achieve 100% Reduction in CPD between Baseline and Month 6 Follow-Up | Month 6
  Verified by exhaled carbon-monoxide (eCO) level.
Percentage of Participants who Achieve 100% Reduction in CPD between End of Intervention (Visit 5) and Month 6 Follow-Up | From Visit 5 (Day 56) up to Month 6
  Verified by exhaled carbon-monoxide (eCO) level.
Change from Baseline in Self-Reported CPD at End of Intervention (Visit 5) | Baseline, Visit 5 (Day 56)
  Verified by exhaled carbon-monoxide (eCO) level.
Change from Baseline in Self-Reported CPD at Month 6 | Baseline, Month 6
  Verified by exhaled carbon-monoxide (eCO) level.
Change from Baseline in Health-Related Quality of Life (HRQOL) Survey Score at End of Intervention (Visit 5) | Baseline, Visit 5 (Day 56)
  8-item self assessment of participants' perceived physical and mental health over time. Each item lists a condition. For each item, participants indicate the number of days the condition applied to them. The total score is the average of responses and ranges from 0-30. Lower scores indicate greater perceived physical and mental health. A reduction in scores indicates perceived physical and mental health improved over the observational period.
Change from Baseline in Health-Related Quality of Life (HRQOL) Survey Score at Month 6 Follow-up | Baseline, Month 6
  8-item self assessment of participants' perceived physical and mental health over time. Each item lists a condition. For each item, participants indicate the number of days the condition applied to them. The total score is the average of responses and ranges from 0-30. Lower scores indicate greater perceived physical and mental health. A reduction in scores indicates perceived physical and mental health improved over the observational period.
Number of Respiratory Symptoms Reported at Baseline | Baseline
Number of Respiratory Symptoms Reported at End of Treatment (Visit 5) | Visit 5 (Day 56)
Number of Respiratory Symptoms Reported at Month 6 Follow-up | Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Omar El-Shahawy, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - NYU Langone Health, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: [Omar.ElShahawy@nyulangone.org]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data and researchers who provide a methodologically sound proposal will be granted access to the data upon reasonable request. Requests should be directed to Omar.ElShahawy@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.